CLINICAL TRIAL: NCT00421005
Title: Safety and Efficacy of Fluvastatin in Heart Transplant Recipients
Brief Title: Fluvastatin After Heart Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Bologna (Other)
Responsible Party: University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 126/2004/U/Sper
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Heart Transplantation; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Fluvastatin

ARMS (2):
- 1 (Experimental): Fluvastatin 80mg
  Interventions: Drug: fluvastatin
- 2 (Active Comparator): Fluvastatin 20, tapered up according to LDL concentration
  Interventions: Drug: fluvastatin

INTERVENTIONS:
Drug: fluvastatin — Fluvastatin 80 mg (Arm 1) vs. Fluvastatin 20 mg (Arm 2) increased according with LDL concentrations
  Other Names: Lescol

SUMMARY:
Statin therapy is a treatment with a proven positive impact on survival after heart transplantation. However, it is unclear whether the beneficial effect of this class of drugs depends solely on their LDL-lowering properties or on anti-inflammatory and immuno-modulatory properties. Thus, this study was designed to compare safety and efficacy of two different strategies: 1. high fixed statin dose vs. 2. low starting dose with LDL-driven doses adjustments.

ELIGIBILITY:
Inclusion Criteria:

* De novo heart transplantation

Exclusion Criteria:

* Known allergy/intolerance to fluvastatin;
* Preexisting neuromuscular disorders;
* Significant liver disease and/or elevation of transaminase exceeding 3 times the ULN
* Severe renal impairment : creatinine > 3 mg/dL
* Intellectual/cognitive impairment likely to compromise informed consent or adherence to protocol or age <18 years.
* Patients refusal
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-11; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Branzi, MD, Study Chair — Alma Mater Studiorum University of Bologna
Locations (1):
- Policlinico S.Orsola-Malpighi, Bologna, Italy

REFERENCES:
- [Background] Kobashigawa JA, Katznelson S, Laks H, Johnson JA, Yeatman L, Wang XM, Chia D, Terasaki PI, Sabad A, Cogert GA, et al. Effect of pravastatin on outcomes after cardiac transplantation. N Engl J Med. 1995 Sep 7;333(10):621-7. doi: 10.1056/NEJM199509073331003. PMID 7637722
- [Background] Holdaas H, Fellstrom B, Cole E, Nyberg G, Olsson AG, Pedersen TR, Madsen S, Gronhagen-Riska C, Neumayer HH, Maes B, Ambuhl P, Hartmann A, Staffler B, Jardine AG; Assessment of LEscol in Renal Transplantation (ALERT) Study Investigators. Long-term cardiac outcomes in renal transplant recipients receiving fluvastatin: the ALERT extension study. Am J Transplant. 2005 Dec;5(12):2929-36. doi: 10.1111/j.1600-6143.2005.01105.x. PMID 16303007
- [Background] Grigioni F, Carigi S, Potena L, Fabbri F, Russo A, Musuraca AC, Coccolo F, Magnani G, Ortolani P, Leone O, Arpesella G, Magelli C, Branzi A. Long-term safety and effectiveness of statins for heart transplant recipients in routine clinical practice. Transplant Proc. 2006 Jun;38(5):1507-10. doi: 10.1016/j.transproceed.2006.02.071. PMID 16797344